CLINICAL TRIAL: NCT04565301
Title: A Comparative Study Between Neostigmine and Dexamethasone as an Adjuvant to Bupivacaine in Adductor Canal Block After Knee Arthroscopy Surgery
Brief Title: Neostigmine and Dexamethasone in Adductor Canal Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Heba Omar Ahmed, Associate professor of Anesthesia, pain management & surgical ICU, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS-161-2020
Record Dates: First submitted 2020-08-26; First posted 2020-09-25 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexamethasone; Calcium Dobesilate; Neostigmine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group C (Placebo Comparator): The patients in this group will be administered 2 ml isotonic saline + 20 ml bupivacaine 0.50 % in the adductor canal block (control group).
  Interventions: Other: NaCl solutions
- Group D (Active Comparator): The patients in this group will be administered 8 mg dexamethasone (2 ml) (23) as adjuvant to 20 ml bupivacaine 0.50 % in the adductor canal block.
  Interventions: Drug: Dexamethasone
- Group N (Active Comparator): The patients in this group will be administered 500 mcg neostigmine (1 ml) + 1 ml isotonic saline (22) as adjuvant to 20 ml bupivacaine 0.50 % in the adductor canal block.
  Interventions: Drug: neostigmine

INTERVENTIONS:
Drug: Dexamethasone — adductor canal block
  Other Names: Decadron
  Arms: Group D
Drug: neostigmine — adductor canal block
  Other Names: prostigmin
  Arms: Group N
Other: NaCl solutions — adductor canal block
  Other Names: normal saline
  Arms: Group C

SUMMARY:
To compare between the efficacy of neostigmine and dexamethasone as an adjuvant to bupivacaine in adductor canal block after knee arthroscopy surgery.

DETAILED DESCRIPTION:
90 participants in this study will be randomized into three groups based on computer generated numbers using computerized generated random tables. The patients enrolled in the study will be transferred to the operation room and monitored all through the surgical procedure using pulse oximeter, non-invasive blood pressure and ECG.

To perform spinal anesthesia ,the patient will be positioned in the sitting position then sterilization of the back using betadine solution 5% will be done then the iliac crest will be identified and the opposite intervertebral space(L4-L5) will be marked then 5 ml of lidocaine 2% will be infiltrated in the skin and subcutaneous tissue then a spinal needle (25G) will be introduced to the intrathecal space and after ensuring that clear cere¬brospinal fluid will be in free flow injection of 15-20mg of bupivacaine 0.5% and 25mcg of fentanyl will be administrated then the patient will be positioned in the supine position.

If hypotension, (decrease in the mean arterial blood pressure of more than 20%from base line) occurs, 9mg intravenous ephedrine will be given with 200ml bolus crystalloids. If bradycardia (heart rate below 50beat / minute) occurs, 0.5mg intravenous atropine will be given. After the surgical procedure the patients will be randomly allocated using computerized generated random tables in to three equal groups and the random numbers will be concealed in closed opaque envelopes which will be kept by the senior anesthesia staff, the three groups are:

* Group neostigmine: The patients in this group will be administered 500 mcg neostigmine (1 ml) + 1 ml isotonic saline (22) as adjuvant to 20 ml bupivacaine 0.50 % in the adductor canal block.
* Group dexamethasone: The patients in this group will be administered 8 mg dexamethasone (2 ml) (23) as adjuvant to 20 ml bupivacaine 0.50 % in the adductor canal block.
* Group control: The patients in this group will be administered 2 ml isotonic saline + 20 ml bupivacaine 0.50 % in the adductor canal block (control group).

With the patient in the supine position, the procedural needle (Braun Stimuplex Ultra Insuflated Echogenic Needle 22G) will be inserted in plane from the anteromedial side at the mid thigh level. It will be advanced through the sartorius muscle and fascia under ultrasound guidance, using a Siemens Acuson X300 ultrasound equipped with a linear transducer after sterilization of the skin with betadine solution 5%, and the adductor canal, with the superficial femoral artery and vein within, will be identified. Once the needle tip will be located in the adductor canal, the anaesthetic solution will be injected anterior to the artery and deep into the sartorius muscle (24) then patient will be transferred to the PACU then to the ward.

Postoperative

1. Postoperative pain will be assessed by visual analog scale (VAS)
2. A fixed dose of intravenous paracetamol 1 gram will be given every 6 hours to all patients in the three groups starting from 1 hour after the ACB.
3. Postoperative pain assessment through VAS will be according to the scale as follow:

   * Pain level 0: no pain
   * Pain level1-3: mild pain
   * Pain level 4-6: moderate pain
   * Pain level 7-10: severe pain
4. Postoperative pain will be managed as follow:

   * Mild pain will be treated with ketolac 30mg IV.
   * Moderate pain will be treated with ketolac 30mg IV + morphine 0.07mg/kg IV.
   * Severe pain will be treated with ketolac 30mg IV & morphine 0.1mg/kg IV. Then patient will be reassessed and recorded as mentioned above and the specific treatment will be repeated after 8 hours from the initial dose according to VAS.
5. Opioids complications such as respiratory depression will be recorded and managed supportively by oxygen mask, controlled airway and if persistent or severe hypoventilation occurs positive pressure ventilation may be needed, nausea and vomiting will be treated with ondansterone (4mg IV).

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing knee arthroscopy surgery.
* Age between 18 years and 65 years.
* Both sexes
* ASA I & ASA II

Exclusion Criteria:

* Patients' refusal
* Allergy to any drug that will be used in the study
* Psychological or mental disorders.
* Disturbance of Conscious level.
* Uncooperative patients
* Coagulopathy
* Contraindications to spinal anaesthesia (e.g.: severe mitral stenosis)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-06-20 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2022-07-27 (Actual)

PRIMARY OUTCOMES:
first rescue analgesia time | 24 hours
  Time (in hours) of first rescue analgesia (morphine) requirement for each group in the first 24 hours following the adductor canal block

SECONDARY OUTCOMES:
morphine consumption | 24 hours
  Total amount of morphine consumed in the first 24 hours following the AC
Visual analogue scale | up to 24 hours
  VAS score at times 0-30 minutes, 1, 2, 4, 8, 12, 18 and 24 hours postoperatively. As visual analouge scale (VAS) is a scale from 0 to 10 where "0" means no pain and "10" means the most severe pain.
sensory block | up to 24 hours
  Duration of sensory block at times 0-30 minutes, 1, 2, 4, 8, 12, 18 and 24 hours postoperatively
Presence of Nausea and vomiting | 24 hours
  through a question answered by yes or no to identify the presence of nausea and vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Heba Omar, Principal Investigator — associate professor of anesthesia and surgical ICU, faculty of medicine, Cairo university
Locations (1):
- Kasr Alainy hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No